CLINICAL TRIAL: NCT02186886
Title: Personalised Medicine: a Break Through Approach for Early Determination of Anti Tumor Necrosis Factor (TNF) Responders and Non Responders Among Patients With Ulcerative Colitis in a Prospective Study With Golimumab (Simponi)
Brief Title: Physiological Intermolecular Modification Spectroscopy (PIMS) in Ulcerative Colitis With Golimumab
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kliniken im Naturpark Altmuehltal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 50831-PIMS-Golimumab-UC
Record Dates: First submitted 2014-07-01; First posted 2014-07-10 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Golimumab; Physiological Intermolecular Modification Spectroscopy; PIMS
MeSH Terms: conditions — Colitis, Ulcerative | interventions — golimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Golimumab (Other): Golimumab: Patients with body weight less than 80 kg initial dose of 200 mg, followed by 100 mg at week 2, then 50 mg every 4 weeks, thereafter // Patients with body weight greater than or equal to 80 kg initial dose of 200 mg, followed by 100 mg at week 2, then 100 mg every 4 weeks, thereafter
  Interventions: Drug: Golimumab

INTERVENTIONS:
Drug: Golimumab — Physiological Intermolecular Modification Spectroscopy

SUMMARY:
Aim of this study is to determine wether the macromolecular spectral characteristic of ulcerative colitis patients - measured by Physiological Intermolecular Modification Spectroscopy (PIMS) - is a predictive factor for response to Simponi treatment

DETAILED DESCRIPTION:
It is widely appreciated that almost all proteins and other biological macromolecular in vivo exist, at least transiently, as components of structural and functional complexes. This transient interaction in simple component solutions have been studied using well established daylight light scattering (LS) method which reflects molecular oscillation (7-12). Protein association, protein unfolding, protein aggregation and cellular crowding are known to affect the normal function of cellular system (13-19). In many cases, the resulting small changes in normal protein-protein intra- and intermolecular interactions are thought to lead to a variety of human diseases (20, 21). Based on these and the acquired knowledge on LS, the cutting edge technology, PIMS has been developed. PIMS is a label free technology that is able to study protein-protein and protein-solvent interactions in multi-component solutions. It provides individual real time dynamic fingerprint of total physiological macromolecular assemblies in a tissue in presence and absence of exogenous molecules (drug or drug candidate, peptide or protein).

This technology is based on dynamic molecular resonance of proteins and macromolecules. Cellular extracts in physiological conditions are frozen at -37°C. Macromolecular spectra are registered as the temperature within the sample raises from -37 to 37°C. This provides, within the organ of interest, dynamic fingerprint of an individual entire macromolecular assemblies. The present technology can therefore rapidly and specifically determine the response of a tissue or cell when an exogenous molecule is administrated. It reflects patient molecular capacity to respond to the drugs effect and allows to identifying different subpopulations within a group in response to a specific treatment. It highlights the responders from non-responders to a given treatment.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe active ulcerative colitis
* qualified for initiating Golimumab therapy, i.e.inadequate response to conventional therapy including corticosteroids and 6-mercaptopurine or azathioprine or intolerance of medical contraindications to such therapies
* must be able and willing to provide written informed consent
* must have a negative tuberculosis screening or if inactive (latent) tuberculosis diagnosed anti-tuberculosis therapy to be started before initiation of Golimumab therapy in accordance with local recommendations

Exclusion Criteria:

* cancer
* type one diabetes
* current infection and/or inflammation other than related to ulcerative colitis
* autoimmune diseases
* any contraindications stated by Golimumab product label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Clinical response | Week 14
  Reduction of partial Mayo Score > 2 points versus baseline

SECONDARY OUTCOMES:
Calprotectin stool levels | Week 6
  Change in calprotectin stool levels at week 6 versus baseline
Calprotectin stool levels | Week 14
  Change in calprotectin stool levels at week 14 versus baseline

OTHER OUTCOMES:
molecular spectral range | Week 14
  Change in molecular spectral ranges versus baseline

CONTACTS AND LOCATIONS:
Overall Officials: Matthias G Breidert, MD, Principal Investigator — Naturpark Kliniken Altmuehltal
Locations (1):
- Kliniken im Naturpark Altmuehltal; Klinik Koesching, Kösching, Germany